CLINICAL TRIAL: NCT04259931
Title: PROSPECTIVE STUDY OF PREDISPOSING FACTORS OF REFRACTARY Clostridium Difficile INFECTION. INFLUENCE OF THE GUT MICROBIOMA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario de Cabuenes (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Hospital Universitario Central de Asturias (Other); Instituto de Productos Lacteos de Asturias (Unknown)
Responsible Party: Principal Investigator, Azucena Rodriguez Guardado, Md PhD, Hospital Universitario de Cabuenes
Other Study IDs: CLOSTRI PROJECT
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; relapse; microbiome
MeSH Terms: conditions — Clostridium Infections; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No relapses: Patients with clostridium difficile infections without relapses
  Interventions: Diagnostic Test: microbiome analysis
- Relapsing patiens: Patients with clostridium difficile infections with relapses
  Interventions: Diagnostic Test: microbiome analysis

INTERVENTIONS:
Diagnostic Test: microbiome analysis — gut microbiome composition of C. difficile infected patients with relapsing (basal, at the end of first treatment, at the begin of the relapses and at four and twelve weeks after definitive treatment) and non-relapsing ( basal and four and twelve week after treatment) , will be analyzed.

SUMMARY:
A higher frequency of recurrences in the University Hospital of Cabueñes (HUCAB) than in other hospitals in our area, including Central University Hospital of Asturias (HUCA) has been found. This increase does not seem to be related to underlying diseases, age, sex or predisposing factors classically described in this type of infection. This high rate of recurrence, together with the absence of response to all conventionally used antibiotic treatments, has important repercussions in the morbidity and mortality of patients, in the ecology of the hospital due to the risk of transmission of a strain of major severity and in the high costs associated with an increase in the hospitalization days of these patients, as well as in an eventual transfer of these to other structures specialized in fecal transplantation.

Two hypotheses are proposed to explain the higher frequency reported:

Hypothesis 1. There are alterations of the microbiome in patients with severe recurrences that favor the appearance of these.

Hypothesis 2. The circulating strain in the hospital has intrinsic characteristics that make it more virulent, such as the presence of virulence or multiresistance factors.

For this reason we design a descriptive, prospective multicentric study that will include all patients older than 18 years diagnosed with C difficile infection at the Central University Hospital of Asturias and the University Hospital of Cabueñes during the year 2020-2021

DETAILED DESCRIPTION:
Clostridium difficile infection (CDI) is currently a priority public health problem. In recent decades, the exponential increase in the incidence and severity of CDI has forced to develop new and better methods of treatment and control of the infection. Currently, it is the most common cause of nosocomial infectious diarrhea, with 20 cases per 100,000 people / year or 15 cases per 1000 hospital discharges.

The identification of risk factors for the CDI has become one of the basic pillars to study in order to improve epidemiological control. Classically known risk factors associated with CDI (hospitalization, advanced age, antibiotic prescription, gastrointestinal surgery) have joined in recent years as a result of recent research (for example, the use of proton pump inhibitors).

One of the main problems offered by the management of the CDI is the role of recurrences. There is no consensus about the definition of recurrence in the international CDI management guidelines, however, it is usually established as the presence of diarrhea in the 30 days after an CDI that had presented positive toxin.

The recurrence of the CDI implies a new level of complexity when dealing with the management of this infection: the recurrence percentages range between 15-50% after an initial episode, establishing in recent studies that it could be reasonable to estimate that 20-25% of the patients will present a recurrence in the first 30 days after finishing the antibiotic treatment for the CDI. In addition, after the first recurrence the risk of presenting a new one increases up to 45%, and the risk of subsequent recurrences doubles after 2 or more recurrences.

The study of recurrence in the CDI is the objective of multiple studies. Its importance is based on both epidemiological and economic reasons, since each episode of recurrence increases hospital costs (in a study carried out by the Spanish Ministry of Health in 2013, it was estimated that each new episode of recurrence entailed an increase in the cost of 1000 euros)

The new lines of recurrence research in CDI try to find associations between severity, microbiome, demographic findings and new risk factors and the possibility of recurrence, in order to try to predict it by developing clinical models predictive of recurrence, which, until now, they only have a very limited role.

Previous data collected by our working group show important differences in the behavior of Clostridium difficile infection between the Central University Hospital of Asturias (HUCA) and the University Hospital of Cabueñes (HUCAB), among which the high number of recurrences and failures to conventional treatments in the latter, being necessary even fecal transplantation as a last therapeutic resource.

In 2017, there were 27 patients with Clostridium difficile infection in the HUCAB, of whom 8 (33.3%) relapsed. In 2018, 4 (22.2%) of 18 patients relapsed, three of them more than three times. Analyzing the characteristics of patients with recurrence within the HUCAB during the years 2017-2018, we found that recurrences are significantly more frequent in patients treated with metronidazole, although this is possibly due to the fact that it is the drug used systematically as the first choice, and diagnosed with hepatopathy without differences between the other treatments, which supports the hypothesis that the differences are due more to the behavior of the strain than to the clinical characteristics of the patients.

A higher frequency of recurrences in the University Hospital of Cabueñes (HUCAB) than in other hospitals in our area, including Central University Hospital of Asturias (HUCA) has been found. This increase does not seem to be related to underlying diseases, age, sex or predisposing factors classically described in this type of infection. This high rate of recurrence, together with the absence of response to all conventionally used antibiotic treatments, has important repercussions in the morbidity and mortality of patients, in the ecology of the hospital due to the risk of transmission of a strain of major severity and in the high costs associated with an increase in the hospitalization days of these patients, as well as in an eventual transfer of these to other structures specialized in fecal transplantation.

Two hypotheses are proposed to explain the higher frequency reported:

Hypothesis 1. There are alterations of the microbiome in patients with severe recurrences that favor the appearance of these.

Hypothesis 2. The circulating strain in the hospital has intrinsic characteristics that make it more virulent, such as the presence of virulence or multiresistance factors We design a descriptive, prospective multicentric study that will include all patients older than 18 years diagnosed with C difficile infection at the Central University Hospital of Asturias and the University Hospital of Cabueñes during the year 2020-2021

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed of C. difficile infection
2. Age older than 18 years old.

Exclusion Criteria:

1. Failing to meet the inclusion criteria
2. If the positive microbiological results were not associated with clinical features of gastrointestinal infection.
3. Patients with incomplete data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We design a descriptive, prospective multicentric study that will include all patients older than 18 years diagnosed with C difficile infeopiction at the Central University Hospital of Asturias and the University Hospital of Cabueñes during the year 2020-2021
  For the purpose of the study we define case as a patient with C. difficile infection demonstrated in stool samples in presence of compatible gastrointestinal diseases.
  We define a positive microbiological result if the patient had a determination of toxin plus GDH positives or there is colonoscopy or histopathological evidence of pseudomembranous colitis. The discordant cases will be confirmed by PCR, and we consider that infection exits if it is positive Recurrence will be considered if the patient presents a new episode of C. difficile infection if he / she presents again compatible clinical and positive microbiological diagnosis in the 60 days following the previous episode.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification of risk factors | 12 weeks
  identify risk factors linked to the appearance of serious relapses in patients infected with Clostridium difficile, with special emphasis on the relationship between changes in the patient's microbiota and the appearance of these recurrences.

SECONDARY OUTCOMES:
Characterization of the circulating strain: profile of resistance, ribotype and presence of virulence factors. | 16 weeks
  Characterization of the circulating strain: profile of resistance, ribotype and presence of virulence factors.
Study of the alterations in the microbiome of Clostridium difficile-infected patients with relapsing and non-relapsing. | six months
  Study of the alterations in the microbiome of Clostridium difficile-infected patients with relapsing and non-relapsing.

CONTACTS AND LOCATIONS:
Overall Officials: Azucena Rodriguez Guardado, MdPhd, Principal Investigator — Hospital Universitario de Cabuenes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradley CW, Burdett H, Holden KL, Holden E, Garvey MI. How do we define recurrence in Clostridium difficile infection? J Hosp Infect. 2019 Jun;102(2):171-173. doi: 10.1016/j.jhin.2018.07.026. Epub 2018 Jul 26. No abstract available. PMID 30055221
- [Background] Pakpour S, Bhanvadia A, Zhu R, Amarnani A, Gibbons SM, Gurry T, Alm EJ, Martello LA. Identifying predictive features of Clostridium difficile infection recurrence before, during, and after primary antibiotic treatment. Microbiome. 2017 Nov 13;5(1):148. doi: 10.1186/s40168-017-0368-1. PMID 29132405
- [Background] Petrosillo N. Tackling the recurrence of Clostridium difficile infection. Med Mal Infect. 2018 Feb;48(1):18-22. doi: 10.1016/j.medmal.2017.10.007. Epub 2018 Jan 12. PMID 29336928
- [Background] Falcone M, Tiseo G, Iraci F, Raponi G, Goldoni P, Delle Rose D, Santino I, Carfagna P, Murri R, Fantoni M, Fontana C, Sanguinetti M, Farcomeni A, Antonelli G, Aceti A, Mastroianni C, Andreoni M, Cauda R, Petrosillo N, Venditti M. Risk factors for recurrence in patients with Clostridium difficile infection due to 027 and non-027 ribotypes. Clin Microbiol Infect. 2019 Apr;25(4):474-480. doi: 10.1016/j.cmi.2018.06.020. Epub 2018 Jun 28. PMID 29964230
- [Background] Song JH, Kim YS. Recurrent Clostridium difficile Infection: Risk Factors, Treatment, and Prevention. Gut Liver. 2019 Jan 15;13(1):16-24. doi: 10.5009/gnl18071. PMID 30400734
- [Background] Ford DC, Schroeder MC, Ince D, Ernst EJ. Cost-effectiveness analysis of initial treatment strategies for mild-to-moderate Clostridium difficile infection in hospitalized patients. Am J Health Syst Pharm. 2018 Aug 1;75(15):1110-1121. doi: 10.2146/ajhp170554. Epub 2018 Jun 14. PMID 29903711
- [Background] Tieu JD, Williams RJ 2nd, Skrepnek GH, Gentry CA. Clinical outcomes of fidaxomicin vs oral vancomycin in recurrent Clostridium difficile infection. J Clin Pharm Ther. 2019 Apr;44(2):220-228. doi: 10.1111/jcpt.12771. Epub 2018 Oct 22. PMID 30350418
- [Background] Asensio A, Bouza E, Grau S, Rubio-Rodriguez D, Rubio-Terres C. [Cost of Clostridium difficile associated diarrhea in Spain]. Rev Esp Salud Publica. 2013 Jan-Feb;87(1):25-33. doi: 10.4321/S1135-57272013000100004. Spanish. PMID 23748655